CLINICAL TRIAL: NCT04518930
Title: Comparing the Effect of High-Fat (Peanuts) Versus High-Protein (Plain Greek Yogurt) Snacks on Appetite Hormones and Satiety Among Overweight and Obese Women
Brief Title: High Fat vs High Protein and Appetite Hormones
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Balqa Applied University (Other)
Collaborators: University of Jordan (Other)
Responsible Party: Principal Investigator, Nahla Bayyari, Clinical professor, Al-Balqa Applied University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HF vs HP-8/2020
Record Dates: First submitted 2020-08-15; First posted 2020-08-19 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Body Weight; Appetitive Behavior; Dietary Exposure; Hormone Deficiency
Keywords: High fat; High protein; Satiety hormones; Appetite; Obesity
MeSH Terms: conditions — Body Weight; Appetitive Behavior; Obesity | interventions — Snacks

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- high fat (Experimental): 26 participants will be provided with (35) g of roasted, not salted peanuts as snack.
  Interventions: Other: Peanuts or plain Greek yogurt
- high protein (Experimental): 26 participants will be provided with (380) g of Plain Greek yogurt after as snack.
  Interventions: Other: Peanuts or plain Greek yogurt

INTERVENTIONS:
Other: Peanuts or plain Greek yogurt — Two different types of dietary snacks
  Other Names: snack

SUMMARY:
This study will investigate the effects of high-protein, high-fat snacks, specifically Greek yogurt, and peanuts, on satiety, gut hormones, and insulin secretion in overweight and obese women. The hypothesis posited that peanuts will exhibit a more beneficial impact on satiety, gut hormones, and insulin levels compared to Greek yogurt. The two-arm parallel randomized trial will involve 52 participants aged 30 to 40 with a BMI between 25-35 kg/m²,and they will be randomly divided into peanut (n=26) and Greek yogurt (n=26) groups. Pre-snack, BMI and dietary intake will be assessed. Appetite sensations will be gauged using a visual analog scale (VAS) upon arrival, and at 30- and 60-minutes post-snack. Pre- and post-snacking, plasma levels of cholecystokinin (CCK), Peptide Tyrosine-Tyrosine (PYY), Glucagon Like Peptide-1 (GLP-1), Ghrelin (GHRL), and insulin will be analyzed.

DETAILED DESCRIPTION:
The study's inclusion criteria will be encompassed women aged between 30 and 40 years, with a body mass index (BMI) ranging from 25 to 35 kg/m². These individuals engaged in light exercise 1-3 times per week (activity factor 1.375) and adhered to a routine of consuming three regular meals, along with two daily snacks, and maintaining a water intake of eight cups and do not have allergies to nuts or yogurt.

All participants should adhere to a 1200 kcal diet plan, which included breakfast, snack 1, lunch, snack 2, and dinner. This diet plan will remain consistent for all participants over a consecutive three-day period, except for the snacks that will be provided during the second visit. The specific snack assigned to each participant will be determined based on a predetermined randomization list. The first experimental group (n=26) will receive a high-protein snack in the form of plain Greek yogurt, while the second experimental group (n=26) will receive a high-fat snack in the form of peanuts.

Prior to intervention, in the first visit all anthropometric and body composition assessments will be performed. On the second visit which will be scheduled after three days of adhering to the 1200 Kcal diet, all participants should arrive at the clinic at 1:00 pm and they should had their breakfast at home at 9:00 am. Upon arrival, a baseline blood samples from each participant will be collected.

At 1:00 pm, participants in the plain Greek yogurt and peanut groups will consume their assigned snacks. Following snack consumption, a validated visual analog scale (VAS) questionnaire will be distributed to assess sensations and appetite levels at 0 minutes (1:00 pm), 30 minutes (1:30 pm), and 60 minutes (2:00 pm).

One hour after their arrival, at 2:00 pm, a second blood sample will be collected from all participants. Serum samples will be used to analyze the Ghrelin, PYY, CCK, Glp-1 and insulin using human ELISA kits.

Statistical analysis will be performed after data entry using the SPSS statistical software. Prior to analysis data will be tested for normality. Descriptive statistics for continuous (means± SD) and categorical variables (frequencies and percentages) along with analytical statistics including t-test for paired and unpaired means and the repeated measures for the general linear model will be performed too. P < 0.05 will consider significant.

ELIGIBILITY:
Inclusion Criteria:

Women aged between 30 and 40 years, with a body mass index (BMI) ranging from 25 to 35 kg/m², engaged in light exercise 1-3 times per week (activity factor 1.375) and adhered to a routine of consuming three regular meals, along with two daily snacks, and maintaining a water intake of eight cups and do not have any allergies, particularly to peanuts, and yogurt.

Exclusion Criteria:

Women aged below 30 years or above 40 years, BMI below 25 kg/m² or above 35 kg/m², engaged in little or no exercise or engaged in moderate to heavy exercise, pregnant or lactating mothers, had allergies to nuts, peanuts, yogurt, milk, or milk products, using medications, hormonal therapy, supplements, oral contraceptives, or herbal/botanical products claimed to suppress appetite. Women in menopausal state, in their menstrual cycle days, or within one week before their menstrual cycle days will be excluded. Those with chronic diseases such as cardiovascular diseases, diabetes, hypertension, kidney diseases, thyroid disorders, gastrointestinal diseases, polycystic ovary syndrome, or androgen disorders, following a weight-reducing diet, experiencing sleep disorders, or sleeping less than 8 hours per day, and consuming less than 8 cups of water per day will also excluded.

Ages: 30 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Overweight and obese females
Enrollment: 52 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2023-10-22 (Actual)

PRIMARY OUTCOMES:
Appetite hormones | one week
  The effects of peanut snacking versus plain Greek yogurt on appetite hormones will be measured on Cholecystokinin, Ghrelin, Peptide YY, and Glucagon Like Peptide-1 and Insulin levels
Appetite sensations | 8 weeks
  The effect of peanut snacking versus plain Greek yogurt on appetite sensations will be measured using validated visual analog scale (VAS) questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Nahla S Al-Bayyari, Ph.D, Study Director — Al-Balqa Applied University
Locations (1):
- Nahla S Al-Bayyari, Salt, Balqa Governorate, Jordan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Al-Bayyari N, Alhameedy M, Omoush R, Ghazzawi H. Exploring the effects of high protein versus high fat snacks on satiety, gut hormones and insulin secretion in women with overweight and obesity: A randomized clinical trial. Obes Pillars. 2025 Sep 27;16:100212. doi: 10.1016/j.obpill.2025.100212. eCollection 2025 Dec. PMID 41079153

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-03-06): https://cdn.clinicaltrials.gov/large-docs/30/NCT04518930/Prot_SAP_000.pdf